CLINICAL TRIAL: NCT07297381
Title: Neuromuscular Electrical Stimulation and Action Observation for Healthy Aging: a Home-based Approach to Promote Sensorimotor Adaptation
Brief Title: Neuromuscular Electrical Stimulation and Action Observation for Healthy Aging
Acronym: PRIN2022
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ambra Bisio (Other)
Collaborators: Universita degli Studi di Genova (Other)
Responsible Party: Sponsor-Investigator, Ambra Bisio, Professor, University of Genova
Organization: University of Genova (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100008-2023-AB-PRIN_Bando2022
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aging, Healthy
Keywords: aging; physical fitness; strength; weight estimation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action Observation - Neuromuscular Electrical Stimulation (Experimental): During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. Meanwhile participants will observe video showing movements of activity of daily living.
  At the end of the warm-up phase, the exercise phase will be administered at functional threshold (the minimum intensity required for a complete arm flexion or at maximal tolerated intensity (f=100Hz, t=400 μs).
  Interventions: Combination Product: Action Observation - Neuromuscular Electrical Stimulation
- Action Observation (Active Comparator): During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. Meanwhile participants will observe video showing movements of activity of daily living.
  At the end of the warm-up phase, participants will receive a NMES sham treatment (f=5Hz, t=100 μs) delivered at sensory threshold, known to be ineffective in increasing muscle strength.
  Interventions: Combination Product: Action Observation
- Neuromuscular electrical stimulation (Active Comparator): During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. Meanwhile participants will observe video showing different landscapes.
  At the end of the warm-up phase, the exercise phase will be administered at functional threshold (the minimum intensity required for a complete arm flexion or at maximal tolerated intensity (f=100Hz, t=400 μs).
  Interventions: Combination Product: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Combination Product: Action Observation - Neuromuscular Electrical Stimulation — During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. Meanwhile participants will observe video showing movements of activity of daily living.
  At the end of the warm-up phase, the exercise phase will be administered at functional threshold (the minimum intensity required for a complete arm flexion or at maximal tolerated intensity (f=100Hz, t=400 μs).
  Arms: Action Observation - Neuromuscular Electrical Stimulation
Combination Product: Action Observation — During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. Meanwhile participants will observe video showing movements of activity of daily living.
  At the end of the warm-up phase, participants will receive a NMES sham treatment (f=5Hz, t=100 μs) delivered at sensory threshold, known to be ineffective in increasing muscle strength.
  Arms: Action Observation
Combination Product: Neuromuscular Electrical Stimulation — During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. Meanwhile participants will observe video showing different landscapes.
  At the end of the warm-up phase, the exercise phase will be administered at functional threshold (the minimum intensity required for a complete arm flexion or at maximal tolerated intensity (f=100Hz, t=400 μs).
  Arms: Neuromuscular electrical stimulation

SUMMARY:
Aging is associated with a decline in muscle strength and the functionality of the perceptual structures involved in proprioception. This decline results in a gradual loss of autonomy in daily activities. Neuromuscular electrical stimulation (NMES) has been shown to be an effective technique in limiting the decline in strength. Action observation (AO) is a cognitive technique, which has been shown to improve motor performance, especially when combined with peripheral stimulation.

The purpose of this study is to evaluate whether a self-administered, home-based intervention combining NMES and AO improves upper limb muscle strength and proprioceptive abilities in healthy elderly individuals.

Participants within the age range of 65-85 years will be recruited for this study. The intervention is scheduled to span a duration of four weeks, encompassing three treatment sessions per week. Participants will be randomly divided into three groups: NMES, AO, and AO-NMES. Assessments will be performed before and immediately after the intervention. They will include muscle strength evaluation (handgrip strength, maximal isometric force of the biceps, bench press power), and perceptual evaluation (weight discrimination during an AO task, weight judgment tasks).

This study may suggest an original approach, cost-effective approach to mitigate the effects of physiological aging on muscle and sensorimotor function, with potential applications for frail populations, unable or unmotivated to perform conventional physical activity.

DETAILED DESCRIPTION:
Aim The purpose of study will be testing the effects of a self-administered, home-based intervention combining NMES and AO for the upper limbs in healthy elderly people on muscle strength and proprioceptive abilities. This will be done by comparing action observation-neuromuscular electrical stimulation (AO-NMES) with action observation (AO) and neuromuscular electrical stimulation (NMES) delivered alone, with the hypothesis that AO-NMES leads to higher improvement than the others. This approach could be a safe, accessible and cost-effective way to maintain or improve neuromuscular function and sensorimotor control in ageing populations. Furthermore, by preserving upper limb function, the intervention could help older adults to retain functional autonomy, reduce their risk of disability and improve their overall quality of life and well-being.

Methods

1. Participants Voluntarily participants will be recruited from the students enrolled in the 'UniGeSenior' program at the University of Genoa. The inclusion criteria are voluntarily participation, age ranges from 65 to 85 years, both male and female, sedentary. Exclusion criteria include neurological or psychiatric disorders, fractures within the past six months, orthopedic or musculoskeletal impairments, uncontrolled hypertension, and regular resistance training (at least once per week), participation in competitive sports.
2. Study design This will be a randomized, double-blind, controlled experimental trial. The study will be registered on ClinicalTrials.gov. The intervention will last four weeks, three sessions per weeks will be performed at home. The intervention will vary according to the assigned group, with all interventions delivered in parallel across the following groups: AO group, NMES group and AO-NMES group. The assignment will be done using the RAND() function in Excel, which generated random numbers that were then used to sort and allocate subjects evenly. During each session, the treatment will last 30 minutes and will include a 10-minutes warm-up phase during which the visual task will be administered, and 20 minutes of exercise phase.

   Before (PRE) and after (POST) the intervention period participant will perform different kinds of assessments (see Evaluation section).
3. Intervention 3.1. Visual stimuli

   The stimuli shown to the participants will change according to the group. In the AO group participants will watch a video showing different instrumental activities of daily living (IADLs), which require considerable force production, executed with the upper limbs by a woman or a man. The IADLs will involve the individual performing the following tasks:
   * Moving a box forward or backward while sitting on a chair
   * Lifting a box onto or bringing it down from a support while standing upright
   * Placing a box onto or removing it from a shelf while standing upright
   * Moving a box from left to right or right to left while sitting on a chair
   * Moving a shopper from right to left or left to right while standing upright
   * Placing a shopper on a shelf or taking it down from a standing position
   * Holding a shopper while remaining upright The same AO task will be proposed to the AO-NMES group. Participants of the NMES group will observe changing landscapes. The visual stimuli will be administered through a tablet (Smartpad 9 Mediacom, Datamatic S.p.A, Milano, Italy) provided to the participants.

   3.2. NMES parameters During the first day of intervention, participant will receive the NMES medical device (I-TECH PHYSIO, IACER srl, Scorzè, Venice, Italy) and will be instructed on how to use it by a researcher expert in sport science.

   During the warm-up phase, the NMES will be set with a frequency of 50 Hz and a pulse duration at 400 μs and the intensity at motor threshold. During the exercise phase, participants in the AO group will receive a NMES sham treatment (f=5Hz, t=100 μs) delivered at sensory threshold, and known to be ineffective in increasing muscle strength. In the NMES and AO-NMES groups, the exercise phase will be administered at functional threshold (the minimum intensity required for a complete arm flexion) or at maximal tolerated intensity (f=100Hz, t=400 μs).
4. Evaluations Experimental evaluations will include strength assessment, weight judgment task and weight discrimination during an AO task. They will be performed on the same day, with appropriate rest periods between each evaluation. One week before the PRE evaluation, in a familiarization session, participants will perform the strength assessment, the familiarization was recommended with elderly people.

Evaluations will be conducted by two researchers with expertise in sport science, who will be blinded to the type of intervention performed by the participants. Possible harms will be recorded non-systematically based on spontaneous reports from participants during the experimental period.

4.1. Strength assessment The aim of this test is to assess the effectiveness of the three interventions in increasing muscle strength and power.

The handgrip strength (kg) of the participants will be assessed with the KERN MAP handgrip dynamometer (KERN & SOHN GmbH). The participants will execute the test standing, with the shoulder adducted, the elbow extended, the forearm and the wrist neutral. They will be required to grip the dynamometer with their maximum strength. The mean value obtained from three repetitions will be considered to assess the right and left handgrip strength. The mean values between left and right handgrip strength will be considered as the outcome parameter of handgrip strength.

During the familiarization session, participants will familiarize with the isometric curl and the bench press test. Regarding the first test, participants perform 10 submaximal repetitions and 3 maximal repetitions. Regarding the second test, they perform two sets of eight to ten repetitions at a submaximal load of bench press, followed by two sets of two repetitions at maximal speed with an empty bar.

During the evaluation, the assessment of biceps maximal isometric force (MIF, N) will be performed using the Chronojump force sensor (Chronojump, Barcelona, Spain) asking participant to perform an elbow flexion. Participants will be assessed from sitting position, holding a bar with both supinated and elbow angle approximately at 90°. The bar will be connected to the force sensor by a static rope. The movement will be executed three times, with 1-minute pause between each repetition. Participants will be instructed to pull as hard as possible to maintain the contraction for at least 2 s with verbal encouragement. The trial with the highest MIF value will be considered as valid. Before the evaluation, a warm-up phase consisting in a set of five repetitions at the loads of 40-60% of the perceived maximum force will be performed.

Bench press test will be executed to assess the force-velocity relationship, and to estimate the maximal power. The test will be preceded by a warm-up consisting of two sets of 10 repetitions at the Smith Machine. During the execution of traditional bench press, participants will stop the bar to the chest for 2 seconds and then will push the bar as fast as possible until the full extension of the elbow. The initial load will be set at 16kg for male and 12kg for female. The load will constantly increase to perform 3-4 sets, number of sets required to obtain an adequate estimate of maximum power, with an execution speed in the last set lower than 0.3 m⋅s- 1. Between each set, 3 minutes of rest will be applied. During this test a linear position transducer will be used (Chronojump, Barcelona, Spain). One end will be attached on the left side of the bar, and the other end will be fixed to the floor. Maximal Power (MP) will be extracted with Chronojump software.

4.2. Weight judgment task The aim of this evaluation is to test the perceived heaviness of an object in a daily life context with the hypothesis that AO-NMES treatment will have positive effect on proprioceptive ability. A point weight judgement task will be performed. The participants will be instructed to judge the weight of a box in kilograms. A one-kilo box will be used for familiarization of the task. Participants will lift the box, positioned in front of them on a table with the handles aligned at hip level, using arm flexion until approximately 45° of flexion is reached. The box used during the weight judgment task will be filled with cast-iron disk, secured to prevent movement, to reach a weight of 4 kg, 7 kg and 10 kg. Participants will not be given information about weights or the number of different weights. Each box will be lifted 5 times. The mean values weight reported by the participant and coefficient of variations will be considered as outcome parameters together with the estimation error computed as the absolute difference between the real and the perceived weight.

4.3. Weight discrimination during an AO task The aim of this test is to evaluate participants' ability to discriminate the weight of an object moved by others during an action observation task. The hypothesis is that by improving both strength and the perception of heaviness, this enhanced ability will transfer to the motor resonance mechanism, thereby assisting participants in accurately evaluating the weight of an object moved by another individual. The weight-discrimination video task is described in a previous paper of our group. Briefly, participants will have to discriminate the weight of two boxes moved in two consecutive actions displayed in a video indicating which is the heaviest box. One of the videos is used as a reference. The weight inside the box in this video is 7 kg. In the other video, the weight inside the box varied from 0 to 15 kg. The number of trials is 112 (16 repetitions for 7 box weight). Just Noticeable Differences (JND), obtained by the psychometric function, will be the outcome parameter.

4.4. Monitoring adherence to the protocol To monitor participants' adherence to the protocol, a researcher will call each participant at the end of every intervention week to ask whether all planned sessions for that week were completed. The reported number of completed sessions will be recorded to support data interpretation.

ELIGIBILITY:
Inclusion Criteria:

* sedenteary peole

Exclusion Criteria:

* neurological or psychiatric disorders
* fractures within the past six months
* orthopedic or musculoskeletal impairments
* uncontrolled hypertension
* regular resistance training (at least once per week)
* participation in competitive sports

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Estimated maximal power | Assessments will be conducted at two time points: (1) baseline (PRE), prior to the start of the intervention, and (2) post-intervention (POST), immediately after completion of the 4-week intervention period
  Power expressed while performing a bench press exercise. This will be evaluated during the "Strength and power assessment "
Maximal isometric strength | Assessments will be conducted at two time points: (1) baseline (PRE), prior to the start of the intervention, and (2) post-intervention (POST), immediately after completion of the 4-week intervention period
  Maximal isometric strength expressed during a isometric curl with the upper limbs. This will be evaluated during "Strength and power assessment "

SECONDARY OUTCOMES:
Error in the estimation of box weigth | Assessments will be conducted at two time points: (1) baseline (PRE), prior to the start of the intervention, and (2) post-intervention (POST), immediately after completion of the 4-week intervention period
  Estimation of the weigth of a box filled with three different weigths. Calculated as the difference between real weigth and participant's response. Ths will be evaluated during "Weight judgment task"
Just noticeble difference (JND) | Assessments will be conducted at two time points: (1) baseline (PRE), prior to the start of the intervention, and (2) post-intervention (POST), immediately after completion of the 4-week intervention period
  JND is the accuracy in discriminating the weigth of two object that are moved by an actor in a video shown to the participants. This will be evaluated during the "Weight discrimination during an AO task"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Genova, Genoa, Liguria, Italy

IPD SHARING:
Plan to Share IPD: No
The focus is not on individual responses, but rather on understanding the effects of the three types of intervention at the group level.

REFERENCES:
- [Background] Albergoni A, Biggio M, Faelli E, Pesce A, Ruggeri P, Avanzino L, Bove M, Bisio A. Sensorimotor expertise influences perceptual weight judgments during observation of a sport-specific gesture. Front Sports Act Living. 2023 Jun 22;5:1148812. doi: 10.3389/fspor.2023.1148812. eCollection 2023. PMID 37426895
- [Background] Albergoni A, Biggio M, Faelli E, Ruggeri P, Avanzino L, Bove M, Bisio A. Aging deteriorates the ability to discriminate the weight of an object during an action observation task. Front Aging Neurosci. 2023 Aug 7;15:1216304. doi: 10.3389/fnagi.2023.1216304. eCollection 2023. PMID 37609031
- [Background] Alcazar J, Guadalupe-Grau A, Garcia-Garcia FJ, Ara I, Alegre LM. Skeletal Muscle Power Measurement in Older People: A Systematic Review of Testing Protocols and Adverse Events. J Gerontol A Biol Sci Med Sci. 2018 Jun 14;73(7):914-924. doi: 10.1093/gerona/glx216. PMID 29309534
- [Background] Alcazar J, Rodriguez-Lopez C, Ara I, Alfaro-Acha A, Manas-Bote A, Guadalupe-Grau A, Garcia-Garcia FJ, Alegre LM. The Force-Velocity Relationship in Older People: Reliability and Validity of a Systematic Procedure. Int J Sports Med. 2017 Dec;38(14):1097-1104. doi: 10.1055/s-0043-119880. Epub 2017 Nov 10. PMID 29126339
- [Background] Iglesias-Soler E, Mayo X, Rial-Vazquez J, Morin-Jimenez A, Aracama A, Guerrero-Moreno JM, Jaric S. Reliability of force-velocity parameters obtained from linear and curvilinear regressions for the bench press and squat exercises. J Sports Sci. 2019 Nov;37(22):2596-2603. doi: 10.1080/02640414.2019.1648993. Epub 2019 Jul 28. PMID 31354059
- [Background] Insausti-Delgado A, Lopez-Larraz E, Omedes J, Ramos-Murguialday A. Intensity and Dose of Neuromuscular Electrical Stimulation Influence Sensorimotor Cortical Excitability. Front Neurosci. 2021 Jan 15;14:593360. doi: 10.3389/fnins.2020.593360. eCollection 2020. PMID 33519355
- [Background] Vivodtzev I, Debigare R, Gagnon P, Mainguy V, Saey D, Dube A, Pare ME, Belanger M, Maltais F. Functional and muscular effects of neuromuscular electrical stimulation in patients with severe COPD: a randomized clinical trial. Chest. 2012 Mar;141(3):716-725. doi: 10.1378/chest.11-0839. Epub 2011 Nov 23. PMID 22116795
- [Background] O'Connor D, Brennan L, Caulfield B. The use of neuromuscular electrical stimulation (NMES) for managing the complications of ageing related to reduced exercise participation. Maturitas. 2018 Jul;113:13-20. doi: 10.1016/j.maturitas.2018.04.009. Epub 2018 Apr 25. PMID 29903643
- [Background] Maffiuletti NA, Gondin J, Place N, Stevens-Lapsley J, Vivodtzev I, Minetto MA. Clinical Use of Neuromuscular Electrical Stimulation for Neuromuscular Rehabilitation: What Are We Overlooking? Arch Phys Med Rehabil. 2018 Apr;99(4):806-812. doi: 10.1016/j.apmr.2017.10.028. Epub 2017 Dec 9. PMID 29233625
- [Background] Langeard A, Bigot L, Chastan N, Gauthier A. Does neuromuscular electrical stimulation training of the lower limb have functional effects on the elderly?: A systematic review. Exp Gerontol. 2017 May;91:88-98. doi: 10.1016/j.exger.2017.02.070. Epub 2017 Feb 17. PMID 28216413
- [Background] Bisio A, Avanzino L, Biggio M, Ruggeri P, Bove M. Motor training and the combination of action observation and peripheral nerve stimulation reciprocally interfere with the plastic changes induced in primary motor cortex excitability. Neuroscience. 2017 Apr 21;348:33-40. doi: 10.1016/j.neuroscience.2017.02.018. Epub 2017 Feb 15. PMID 28214579
- [Background] Bisio A, Avanzino L, Lagravinese G, Biggio M, Ruggeri P, Bove M. Spontaneous movement tempo can be influenced by combining action observation and somatosensory stimulation. Front Behav Neurosci. 2015 Aug 21;9:228. doi: 10.3389/fnbeh.2015.00228. eCollection 2015. PMID 26441565
- [Background] Bisio A, Avanzino L, Gueugneau N, Pozzo T, Ruggeri P, Bove M. Observing and perceiving: A combined approach to induce plasticity in human motor cortex. Clin Neurophysiol. 2015 Jun;126(6):1212-1220. doi: 10.1016/j.clinph.2014.08.024. Epub 2014 Oct 2. PMID 25454343